CLINICAL TRIAL: NCT02253030
Title: Optical Coherence Tomography Angiography in Neovascular Age-related Macular Degeneration
Brief Title: OCT Angiography in Wet AMD
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Steven Bailey, MD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: IRB#000010535
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration (AMD)
Keywords: AMD; OCT; Angiography; Macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Newly-diagnosed, untreated wet AMD: This group will be adults newly diagnosed with wet AMD who have not undergone any treatment for the condition. Their data will be gathered only once, prior to treatment.
  Interventions: Device: Optical Coherence Tomography
- Wet AMD undergoing "as-needed" treatment: This group will be adults undergoing treatment as-needed for wet AMD. They will be followed monthly over the course of 1 year.
  Interventions: Device: Optical Coherence Tomography
- High-risk eyes: This group will be adults with wet AMD in one eye and findings of dry AMD in the other. The eye with dry AMD will be followed every 6 months for 3 years.
  Interventions: Device: Optical Coherence Tomography
- Wet AMD undergoing a "treat and extend" strategy: This group will be adults with wet AMD undergoing treatment under the "treat and extend" strategy. (The "treat and extend" strategy increases the intervals between treatments as long as the macula remains dry.) They will be followed over the course of 1 year with extra imaging before extending follow-up intervals.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography

SUMMARY:
The primary goals of this study are to use optical coherence tomography (OCT) angiography (blood vessel mapping) to:

1. diagnose the presence of new blood vessels in wet age-related macular degeneration (AMD)
2. evaluate patients undergoing treatment for wet AMD
3. determine if reduced flow to the choroid is a risk factor for developing wet AMD.

ELIGIBILITY:
Inclusion Criteria (Groups with wet AMD):

* Adults aged 50 and older with clinical findings of treatment-naïve (never treated) neovascular AMD with active new blood vessel growth confirmed by clinical testing will be considered

Inclusion Criteria (Group with healthy eyes)

* No evidence of retinal disease
* Refractive error greater than +3.00 diopters or -7.00 diopters (glasses Rx)
* No recent eye surgery in the last 4 months
* No significant cataract to interfere with the quality of the imaging

Exclusion Criteria (All Groups):

* Inability to give informed consent
* Significant kidney disease
* Blood pressure greater than 180/110
* Previous macular laser treatment
* Inability to maintain stable fixation during OCT imaging
* Visual acuity worse than 20/200

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both female and male participants over the age of 50 are being studied.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2014-09; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measure of choroidal neovascular (CNV) vessel area in mm2 | 1 year
Measure of CNV membrane area in mm2 | 1 year
Measure of CNV length density in mm | 1 year
Measure of retinal fluid volume in mm3 | 1 year
Measure of drusen area in mm2 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Bailey, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Casey Eye Institute, Oregon Health & Science University, Portland, Oregon, United States